CLINICAL TRIAL: NCT05860660
Title: Assessment of Screen Use and Impact of Excessive Smartphone Use on Adult Health
Brief Title: Screens, Virtual Reality and Digital Addiction (EVADD)
Acronym: EVADD
Status: Completed | Type: Observational
Sponsor: Institut Rafael (Other)
Responsible Party: Sponsor
Other Study IDs: IR-2023/0001; 2023-A00312-43 (Other: National Agency for the Safety of Medicines and Health Products (ANSM, France))
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-07

CONDITIONS: Internet Addiction Disorder
Keywords: Smartphone; Social Media
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: survey — questionnaires

SUMMARY:
This is an observational study questionnaire-based. This study will be carried out to evaluate the methods of consumption (work/outside work), the characteristics of the tools used, the addictive risk, the consequences on mental and physical health and the impact on quality of life of people exposed to screens and smartphones.

A sample of 800 000 people will be used to learn about the entire French population. Participants will be asked to respond to an anonymous digital survey.

The ultimate goal of this work is to have quality information to help facilitate therapeutic efforts in support of those who may need it.

DETAILED DESCRIPTION:
Inappropriate use of the smartphone is defined as excessive use of the technological tool interfering with social and/or professional activities causing negative consequences such as the alteration of certain cognitive functions such as attention. In addition, the excessive use of smartphones has generated a new form of digital symptoms such as NOMO or nomophobia (addiction to mobile phones by compulsive checking of new messages or social networks) and FOMO (fear of being excluded enriching social experiences, Fear of Missing Out).

From the perspective of social media addiction, research has shown that there is a fine line between habitual, frequent, unproblematic use and problematic and possibly addictive use of social media. Users who express symptoms and consequences traditionally associated with substance addiction (salience, mood changes, tolerance phenomenon, craving, withdrawal, relapse) could be addicted to social media.

Nowadays, abstinence from digital media and consumption cannot realistically be achieved in the context of SR addiction, as the internet and social media have become essential parts of our lives. Rather than shutting down social media altogether, therapy should focus on establishing controlled social media use and digital media awareness.

This study will be carried out to evaluate the methods of consumption (work/outside work), the characteristics of the tools used, the addictive risk, the consequences on mental and physical health and the impact on quality of life of people exposed to screens and smartphones.

A sample of 800 000 people will be used to learn about the entire French population. Participants will be asked to respond to an anonymous digital survey.

This is an observational study questionnaire-based. The ultimate goal of this work is not to overpathologize daily behaviours, but to have quality information to help facilitate therapeutic efforts in support of those who may need it.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older (adult)
* members of the PRO-BTP insurance (email list)
* understanding French language

Exclusion Criteria:

* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French population, adults, liste of members of the PRO-BTP insurance, volunteers
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
percentage of participants with addictive behaviour | 6 months
  Percentage (%) of participants with more than 5 positive answers (YES) in the Smartphone Questionnaire containing 15 questions which suggests addictive behaviour

SECONDARY OUTCOMES:
percentage of participants using video games | 6 months
  Percentage (%) of participants who answered YES to the use of video games and analysis of the "Gaming Disorder-20 items" questionnaire from a scale of 1 (strongly disagree) to 5 (strongly agree)
Percentage of participants using online gambling | 6 months
  Percentage (%) of participants who answered YES to the use online gambling and and analysis of the "online gambling - 9 items" questionnaire on a scale of 0 to 3 (0: Never, 1: Sometimes, 2: Most of the time, 3
Percentage of participants using social media networks | 6 months
  Percentage (%) of participants who answered YES to the various questions on social networks , and analysis of the questionnaire "time spent on social media networks"

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Rafael, Levallois-Perret, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided